CLINICAL TRIAL: NCT01290783
Title: Randomized Double-blind Phase III Trial of FOLF(HA)Iri vs FOLFIRI for Second or Third Line Therapy in Irinotecan-naïve Patients With Metastatic Colorectal Cancer
Brief Title: Trial of FOLF(HA)Iri Versus FOLFIRI in mCRC
Acronym: FOLF(HA)iri
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alchemia Oncology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACO-002
Record Dates: First submitted 2011-01-31; First posted 2011-02-07 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2014-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC; CRC; colorectal; irinotecan; Hyaluronic acid; Hyaluronan
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFIRI (Active Comparator)
  Interventions: Drug: Irintoecan
- FOLF(HA)iri (Experimental)
  Interventions: Drug: HA-Irinotecan solution for Infusion

INTERVENTIONS:
Drug: Irintoecan — * Irinotecan, 180 mg/m2 IV, over 90 minutes, day 1 (in patients > 75 years of age, the irinotecan dose in must be reduced to 150 mg/m2).
  * Leucovorin, 400 mg/m2, or levoleucovorin, 200 mg/m2, IV over 90 minutes with irinotecan.
  * 5-FU, 400 mg/m2 IV bolus day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion.
  * Repeat every two weeks.
  * 8 months of treatment.
  Arms: FOLFIRI
Drug: HA-Irinotecan solution for Infusion — * HA-Irinotecan (irinotecan 180 mg/m2), IV, over 90 minutes, day 1 (in patients > 75 years of age, the irinotecan dose in must be reduced to 150 mg/m2).
  * Leucovorin, 400 mg/m2, or levoleucovorin, 200 mg/m2, IV over 90 minutes with irinotecan.
  * 5-FU, 400 mg/m2 IV bolus day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion.
  * Repeat every two weeks
  * 8 months of treatment.
  Arms: FOLF(HA)iri

SUMMARY:
Trial design:

* Phase III, FOLFIRI versus FOLF(HA)iri (the FOLFIRI regimen with "Hyaluronic acid-Irinotecan" or "HA-Irinotecan") regimen.
* Patients with mCRC (metastatic colorectal cancer), 2nd/3rd line irinotecan naïve.
* Randomized 1:1, double-blinded, multi-centre, multi-national (Australia, Bulgaria, Poland, Serbia, Russia, Ukraine and the United Kingdom).
* Dosing regimen:

  * Irinotecan (180 mg/m2) or HA-Irinotecan (180 mg/m2), IV, over 90 minutes, day 1 (in patients > 75 years of age, the irinotecan and HA-Irinotecan dose in must be reduced to 150 mg/m2).
  * Leucovorin, 400 mg/m2, or levoleucovorin, 200 mg/m2, IV over 90 minutes with irinotecan.
  * 5-fluorouracil (5-FU), 400 mg/m2 IV bolus day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion.
  * Repeat every 2 weeks for 8 months.
* Patient accrual over approximately 12-14 months.
* Monitoring to 18 months post-randomization.
* 390 patients.
* Progression Free Survival (PFS) primary endpoint.
* Safety analysis on the initial 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer with disease progression after first or second line chemotherapy
* Irinotecan naïve.
* ECOG performance status of 0 or 1.
* Measurable disease, i.e. at least one measurable metastatic lesion (spiral CT or MRI).
* Histological proof of colorectal cancer.
* 18 years of age and older.
* Adequately recovered from and at least 4 weeks after recent surgery or chemotherapy.
* Women of child-bearing potential (WOCBP) and male partners of WOCBP must agree to use adequate contraception.
* Patient consent obtained and signed according to local and/or national ethics.
* CT or MRI scan of chest/abdomen/pelvis within 21 days prior to randomization.
* Hematology done within 14 days prior to randomization.
* Chemistry done within 14 days prior to randomization.

Exclusion Criteria:

* History of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for > 5 years.
* Locally advanced or recurrent disease only.
* Unsuitability for irinotecan including known Gilbert's syndrome, active inflammatory bowel disease or chronic diarrhea greater than or equal to grade 2.
* Abdominal or pelvic radiation therapy within the last 12 months.
* Women who are pregnant or breastfeeding.
* Any condition (e.g., psychological, geographical) that would render the protocol treatment dangerous.
* Significant cardiac disease.
* Untreated or symptomatic brain or central nervous system (CNS).
* Presence of pleural effusion or ascites requiring therapeutic thoracocentesis or paracentesis.
* Current partial or complete bowel obstruction.
* Concomitant active infection.
* Enrolled in any other investigational trial, unless treatment in that trial has been discontinued at least 30 days prior to signing the Informed Consent for the ACO-002 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 20 months

SECONDARY OUTCOMES:
Safety | After initial 20 patients receive 2 cycles, then 6 monthly thereafter.
  Diarrhea and haematology

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gibbs, MD, Principal Investigator — Melbourne Health
Locations (5):
- Australia (5):
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Western General Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Border Medical Oncology, Wodonga, Victoria

REFERENCES:
- [Background] Gibbs P, Clingan PR, Ganju V, Strickland AH, Wong SS, Tebbutt NC, Underhill CR, Fox RM, Clavant SP, Leung J, Pho M, Brown TJ. Hyaluronan-Irinotecan improves progression-free survival in 5-fluorouracil refractory patients with metastatic colorectal cancer: a randomized phase II trial. Cancer Chemother Pharmacol. 2011 Jan;67(1):153-63. doi: 10.1007/s00280-010-1303-3. Epub 2010 Mar 24. PMID 20333384